CLINICAL TRIAL: NCT03862508
Title: Efficiency of Plyometric Work Together With the Use of Ballast Weight in Lower Limbs in the Improvement of Performance in Jumpers From 18 to 40 Years Old. Nonrandomized Pilot Study.
Brief Title: Plyometric Work Together With the Use of Ballast Weight in Lower Limbs in the Improvement of Performance in Jumpers
Acronym: PLIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PLIO project
Record Dates: First submitted 2019-02-27; First posted 2019-03-05 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Athletes
Keywords: Jump; Plyometrics; Training; Performance; Powerinstep; Non-randomized clinical trial
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Five Plyometric exercises
  Interventions: Other: Plyometric exercises
- Control (No Intervention): Subjects included in the control group will not receive any intervention

INTERVENTIONS:
Other: Plyometric exercises — Jump Drop Jump, dropping the subject from a height of 30cm and then make a vertical jump.
  Long jumps asking the athletes to take momentum and make a leap forward trying to reach the greatest possible distance.
  Jump Countermovement jump unilaterally, alternating the lower extremities. Jumps 180º with the athletes maintaining a semi-squat position. Jump Countermovement jump repeatedly starting from an upright position and the upper extremities in both hips.
  All the exercises will be done through 8 repetitions per session during the first two weeks, increasing two repetitions every two weeks (until reaching 12 repetitions at the end of the intervention).
  For the realization of each one of the exercises, the ballasted weight will be used (Powerinstep® model).
  Other Names: Plyometric training programme with Powerinstep
  Arms: Experimental

SUMMARY:
Introduction. The high jump is a discipline that use the shortening-stretching cycle. Plyometric exersices emply an eccentric load followed by concentric contraction. Powerinstep is a tool training by means of weigthed weigth whose objective is improving performance in athletes.

Aim. Evaluate efficacy of plyometric training with Powerinstep® in lower limbs, in the performance improvement in professional height jumpers from 18 to 40 years old.

Study design. Non-randomized clinical trial, single bind, with follow-up period.

Methods. 20 athletes will be recruited, that will be randomized to the two study groups: experimental (they carry out a plyometric training programme with Powerinstep) and control (won't be made a intervention on the subjects included in this group). The intervention consists of 6 week, with 2 session for week of 15 minutes duration each. The dependent variables will be the height of the jump, the time of flight, the reaction speed and the impulse force, measures though a pressure platform (model T-PLATE), employing Countermovement Jump, Abalakov and Drop Jump tests. We will make a descriptive statistical analysis. The Shapiro-Wilk statistical test will be used to calculate normality. Trough t-student test of repeated measures and an ANOVA of repeated measures will be calculated the difference between distinct assessment (preintervention, postintervention and follow-up) and the effect intra and inter subject, respectively.

Expected results. We want to observe the changes in performance improvement in height jumpers.

ELIGIBILITY:
Inclusion Criteria:

* Height jumpers
* Age between 18 and 40 years
* Currently participate in the competitive field

Exclusion Criteria:

* Present medical diagnosis of musculoskeletal pathology
* Who have not had musculoskeletal injuries in the last month
* Not signed the informed consent document.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline jump height after intervenion and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The height of the jump will be measured on the Countermovement Jump test. The evaluating physiotherapist will stand in front of the subject, who will start from an upright position with the arms on both hips, and will go to a position of flexion of lower members at 90º. Finally, we will ask the subject for a vertical jump on the pressure platform. The results of this test are measured in centimeters and the higher the score, the greater the vertical jump capacity.

SECONDARY OUTCOMES:
Change from baseline impulse force after intervention and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The impulse force will be measured with the Abalakov test. The evaluator will be placed in front of the evaluated, previously in an upright position, asking him to go to a position of flexion of lower limbs of 90º and then, assisted by the impulse of the arms, perform a jump on the pressure platform. The unit of measurement of the results of this test is the Newton, indicating a higher score indicates a greater impulse of the jump.
Change from baseline vertical jump after intervention and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The vertical jump will be measured with the Drop Jump test. In this test, the physiotherapist will stand in front of the subject, who in an upright position will be dropped from a height of 30 centimeters on the pressure platform, then performing a vertical jump with the help of the arms. The results, in this test, are measured in centimeters, where a higher score indicates a greater vertical jump.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain

IPD SHARING:
Plan to Share IPD: No